CLINICAL TRIAL: NCT00749307
Title: Effects of Supplementation With Algal Triacylglycerols Versus Placebo on Heart Rate Variability in Elderly Patients
Brief Title: Effects of Docosahexaenoic Acid (DHA) on Heart Rate Variability in Elderly Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: IRCCS San Raffaele (Other); DSM Nutritional Products, Inc. (Industry); Pharmanutra s.r.l. (Unknown)
Responsible Party: Francesco Maria Serino, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ALFAHRV01; EudraCT number 2008-005715-18
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Arrhythmia
Keywords: Heart rate variability; Docosahexaenoic acid; DHA; Long chain fatty acids; Long chain polyunsaturated fatty acids; Algal fatty acids; Schizochytrium; Omega 3; Death, Sudden, Cardiac; Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac; Death, Sudden, Cardiac | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA)
  Arms: 1
Dietary Supplement: Placebo
  Arms: 2

SUMMARY:
The purpose of this study is to test the hypothesis that dietary supplementation with an algal source of docosahexaenoic acid (DHA) can improve the heart rate variability in elderly patients.

DETAILED DESCRIPTION:
In western countries, sudden cardiac death (SCD) represents the most common form of cardiovascular death. SCD is often caused by ventricular arrhythmias in patients with a known history of ischemic heart disease but it may also occurs in healthy persons.

In the last years has been extensively studied the protective role of long-chain n-3 polyunsaturated fatty acids (n-3 LCPUFA) against SCD both in healthy persons and in patients affected by coronary artery disease.

The hypothesis that these evidences could be ascribed to an antiarrhythmic effect of n-3 LCPUFA, has been corroborated by the observation of a direct relationship between the dietary intake of these nutrients and a better cardiac autonomic control.

This pathway, in particular, has been confirmed by the analysis of changes in heart rate variability.

Most studies in this field used n-3 LCPUFA derived from fish oil, composed by a combination of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). At our knowledge there are few studies available evaluating the isolated role of DHA, derived from alternative sources of n-3 LCPUFA, as the microalgae, in the prevention of fatal arrhythmias.

ELIGIBILITY:
Inclusion Criteria:

* Age above 65 years

Exclusion Criteria:

* Treatment with or allergy to polyunsaturated fatty acids
* Diagnosis of arrhythmia or antiarrhythmic therapy
* Anticoagulant therapy (except acetylsalicylic acid)
* Pacemaker
* Bleeding diathesis
* Recent cerebral hemorrhage (less than 6 months)
* Thyroid dysfunction

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Heart rate variability (HRV) | basal - 12 weeks - 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele Antonelli Incalzi, MD, Study Director — Campus Bio-Medico University; Giuseppe Rosano, MD, Study Director — IRCCS San Raffaele Pisana. Department of Medical Sciences. Cardiovascular Research Unit.; Francesco M Serino, MD, Principal Investigator — Campus Bio-Medico University; Marco Miceli, MD, Principal Investigator — IRCCS San Raffaele Pisana. Department of Sciences. Cardiovascular Research Unit.
Locations (1):
- IRCCS San Raffaele Pisana. Department of Medical Sciences. Cardiovascular Research Unit., Rome, RM, Italy